CLINICAL TRIAL: NCT03631225
Title: Vectra InVolved Informed Decision Outcome Study (VIVID): A Prospective Randomized Controlled Trial Evaluating the Effect of Guided Care With Vectra Compared to Treatment as Usual in Patients With Rheumatoid Arthritis
Brief Title: The Effect of Guided Care With Vectra Compared to Treatment as Usual in Patients With Rheumatoid Arthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Other Study IDs: 133-CL-01
Record Dates: First submitted 2018-08-03; First posted 2018-08-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Vectra; Radiographic Projections
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Guided-Care Arm: Physicians will use the reported Vectra score to guide treatment decisions
  Interventions: Diagnostic Test: Vectra
- Usual Care Arm: Physicians will treat patient per standard of care without the use of the Vectra score

INTERVENTIONS:
Diagnostic Test: Vectra — Each arm will have the Vectra test however, scores will not be provided for the Usual Care Arm until end of study (12 month time point)
  Groups: Guided-Care Arm

SUMMARY:
The goal of treating patients diagnosed with rheumatoid arthritis (RA) is to achieve remission or low disease activity and thereby prevent joint damage, loss of physical function, and disability. Optimal management requires regular assessment of disease activity, with treatment changes made as needed for optimal efficacy. Vectra is a blood serum test that looks at 12 biomarkers and produces a score on a scale of 1 to 100. The Vectra score has been shown to be the strongest predictor of risk for progression of disease. There is opportunity to gain more information about the utility of Vectra in a real-world clinical setting. This study will, therefore, evaluate the utility of Vectra for guiding treatment decisions and improving RA-related outcomes in comparison with usual care, which will not include Vectra testing. This study will enable a direct evaluation of the clinical benefit associated with using Vectra to guide treatment decisions in patients with RA.

DETAILED DESCRIPTION:
Disease activity in RA can be assessed by physical examination, patient-reported outcomes (PROs) or laboratory tests. Joints counts and PROs are partly or entirely subjective. Their ability to support clinical assessment is limited in certain settings, including for RA patients with common comorbidities, such fibromyalgia, obesity, or depression, or with clinically uncertain inflammatory burden. It can be difficult to assess the origin of ongoing pain in such patients using clinical assessment alone. The two blood tests routinely used to assess RA disease activity, erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP), are objective but are in the normal range in more than half of RA patients with active disease, which reduces their negative predictive value and greatly limits their utility. These clinical and laboratory measures are variously combined in composite scores of RA disease activity, such as the 28-joint count Disease Activity Score (DAS28) or the Clinical Disease Activity Index (CDAI) which are not widely used in the US outside of clinical trials because complete, formal joint counts are time-consuming and composite scores pose logistic challenges in a busy clinic setting.

Radiographic progression (RP) is a validated endpoint accepted by the FDA for clinical trials that reflects RA-related damage to joints. It is associated with long-term disability. Optimal care requires that the risk of progression be reduced. Quantitative scoring of RP is performed only for clinical trials and is not used for assessing RP risk in clinical practice. Rheumatologists are generally not trained to score radiographs and they are very time-consuming to score, typically taking 20 or more minutes per patient for a skilled reader. However, they are a valuable scientific endpoint in that they serve as a valid proxy for long term damage and associated RA-related disability. Conventional clinical and laboratory-based measures of RA disease activity are weak predictors of RP, including among patients in clinical remission, where progression can still occur. Thus, an objective, convenient measure that reflects pathologically meaningful disease activity and predicts risk for progression is needed for optimal management of RA.

The multi-biomarker disease activity (MBDA) test, Vectra®, is an objective tool that combines serum concentrations of 12 biomarkers in a validated algorithm to produce a score on a scale of 1 to 100. The MBDA test was subsequently adjusted to account for the effects of age, sex, and leptin (a surrogate for adiposity) in patients with rheumatoid arthritis (RA). The Vectra score has been shown to be the strongest predictor of risk for RP, compared with conventional disease activity measures, including DAS28-CRP, CRP and the swollen joint count. In multivariate analyses, it was the only disease activity measure to independently predict RP. High Vectra scores (>44) are associated with greatest risk for progression and low and moderate scores with very low risk. Across multiple studies, Vectra has a negative predictive value for progression of 93-97%, and in a meta-analysis, the relative risk for progression with a high Vectra score (5.1) is substantially greater than with a high DAS28-CRP (1.4) or high CRP (1.6). The predictive value of Vectra exists even when the Vectra score and clinical measures are discordant, which means that patients with high DAS28-CRP have little risk for RP when Vectra score is low and, conversely, patients with low DAS28-CRP have high risk for RP when Vectra score is high.

Thus, reducing high Vectra scores should be a primary goal of therapy, regardless of the level of clinical disease activity, and using Vectra scores to guide therapy should be an effective way to prevent radiographic progression. A recent prospective study of daily and diurnal variation in Vectra score established that the minimally important difference (MID) in Vectra score - i.e., the magnitude of change in Vectra score that is needed to be confident that it reflects real biologic change and is not due only to random variation - is greater than or equal to 8 Vectra units. Accordingly, a threshold of 8 can be used in guidances for using Vectra to evaluate treatment response.

The primary objective is to compare the clinical response from baseline to 12 months among patients with RA receiving Vectra-Guided care versus those receiving usual care.

The secondary objectives of this study are to:

* Evaluate the rate of radiographic progression from baseline to year 1 among patients with RA whose care is guided by Vectra relative to those receiving usual care.
* Evaluate changes in Vectra score from baseline to 6 months and baseline to year 1 among patients with RA whose care is guided by Vectra DA relative to those receiving usual care.
* Evaluate clinical response from baseline to 1 year among patients with RA receiving Vectra-guided care relative to those receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old at screening visit
* Diagnosed with RA according to 1987 or 2010 criteria of the American College of Rheumatology
* At the time of the pre-baseline visit, patient has a CDAI score of >10
* Currently taking one or more non-biologic or biologic DMARD at screening and for at least the 3 months prior to screening
* Visit at time of screening scheduled as part of routine care
* Subject and/or physician willing to consider treatment change at screening
* No expectation of imminent treatment change at screening or baseline visit

Exclusion Criteria:

* Currently taking an anti-IL-6R drug (tocilizumab, sarilumab)
* Any contraindication, administrative barrier, or financial limitation (e.g. no insurance coverage) that makes it impossible for subject to receive at least one new biologic or JAKi therapy for RA
* Active infection
* History of malignancy within the past 5 years or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ that has been treated or excised in a curative procedure
* Current enrollment in another clinical trial
* Any condition or circumstance that makes it likely the patient will not be able to complete the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with active rheumatoid arthritis at pre-determined clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
ACR20 response at 12 months | Baseline visit to 12 months
  The primary endpoint of this study is ACR20 response, as compared between the guided-care arm and the usual care arm using a generalized estimating equation for logistic regression at six months that accounts for differences in baseline risk factors between the two arms and intracluster correlation induced by site cluster randomization.

SECONDARY OUTCOMES:
Radiographic progression at 1 year | Baseline to 12 months (1 year)
  A secondary endpoint of this study is the rate of radiographic progression at 1 year, as measured by the change (Δ) in modified total Sharp score (mTSS) from baseline to 1 year.
Change in Vectra score | Baseline to 6 months, and baseline and 12 months (1 year)
  Another secondary endpoint of this study is the change in Vectra score.
ACR20 response at 6 months | Baseline to 12 months (1 year)
  Another secondary endpoint of this study is ACR20 response, as compared between the guided-care arm and the usual care arm using a generalized estimating equation for logistic regression at 12 months (1 year) that accounts for differences in baseline risk factors between the two arms and intracluster correlation induced by site cluster randomization.

OTHER OUTCOMES:
Exploring a change in the definition of non-progression less than or equal to 5 | Baseline to 12 months (1 year)
  The percentage of patients with radiographic non-progression, defined as ΔmTSS less than or equal to 5 from baseline to 1 year.
Exploring a change in the definition of non-progression less than or equal to 3 | Baseline to 12 months (1 year)
  The percentage of patients with radiographic non-progression, defined as ΔmTSS less than or equal to 3 from baseline to 1 year.
Change in physical function measured by HAQ-D1 | Baseline to 12 months (1 year)
  Change in physical function measured by the Health Assessment Questionnaire Disability Index (HAQ-DI)
Change in clinical disease activity measured by Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline to 12 months (1 year)
  Change in clinical disease activity measured by PROMIS (Fatigue, Pain Interference, and Social Participation).PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions.
Change in physical function measured by PROMIS | Baseline to 12 months (1 year)
  Change in physical function measured by the Patient Reported Outcomes Measurement Information System (PROMIS) physical function 10 (PF10). PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions.
Change in clinical disease activity measured by RAPID3 | Baseline to 12 months (1 year)
  Change in clinical disease activity measured by Routine Assessment of Patient Index Data 3 (RAPID3)
Change in clinical disease activity measured by CDAI | Baseline to 12 months (1 year)
  Change in clinical disease activity measured by the Clinical Disease Activity Index (CDAI)
Change in clinical disease activity measured by SDAI | Baseline to 12 months (1 year)
  Change in clinical disease activity measured by the Simplified Disease Activity Index (SDAI)
Change in clinical disease activity measured by DAS28-CRP | Baseline to 12 months (1 year)
  Change in clinical disease activity measured by the Disease Activity Score 28-joint count C reactive protein (DAS28-CRP)
The frequency of changes in RA medications [non-biologic, biologic, or targeted synthetic disease modifying anti-rheumatic drugs (DMARDs)] | Baseline to 12 months (1 year)
  Defined as the number of changes per subject per year in type or dosage of prescribed RA medication during the study period.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Bio Solutions Clinical Research, La Mesa, California
  - Brigid Freyne, MD, Murrieta, California
  - J. Lee MD Medical Corp, Orange, California
  - Delaware Arthritis, Lewes, Delaware
  - AARDS Research, Inc., Aventura, Florida
  - Robert W. Levin, MD, PA, Clearwater, Florida
  - Artemisa Analytics, Miami, Florida
  - Rheumatology Associates of Central Florida, P.A., Orlando, Florida
  - Clin-Med Research & Development, LLC, South Miami, Florida
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Clinvest Research, LLC., Springfield, Missouri
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Southern Ohio Rheumatology Inc., Wheelersburg, Ohio
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, PC, Wexford, Pennsylvania
  - PA Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Accurate Clinical Research, Baytown, Texas
  - Pioneer Research Solutions, Inc, Cypress, Texas
  - Accurate Clinical Research, Houston, Texas
  - CardioVoyage, Sherman, Texas
  - Center for Arthritis and Rheumatic Diseases, P.C., Chesapeake, Virginia
  - Arthritis and Osteoporosis Center of Northern Virginia, Manassas, Virginia
  - Center for Arthritis and Rheumatic Diseases., P.C., Suffolk, Virginia
  - Arthritis Northwest, PLLC, Spokane, Washington
  - Aurora Rheumatology and Immunotherapy Center, Franklin, Wisconsin

IPD SHARING:
Plan to Share IPD: No